CLINICAL TRIAL: NCT07032987
Title: Optimising Analgosedation in Extracorporeal Membrane Oxygenation (ECMO) Using a Co-designed Analgosedation Protocol
Brief Title: Improving Sedation Practice in Critically Ill Adult Patients Using a Co-designed Sedation Protocol
Acronym: ECMO-SED
Status: Not yet recruiting | Type: Observational
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: IRAS number: 332457
Record Dates: First submitted 2025-06-09; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-05

CONDITIONS: Intensive Care Medicine; Respiratory Distress Syndrome (RDS); Sedation and Analgesia; ExtraCorporeal Membrane Oxygenation (ECMO); Sedation for Mechanical Ventilation; Cardiogenic Shock; Opioid Analgesia; Analgesia
Keywords: extracorporeal membrane oxygenation; sedation; opioid; sedatives; analgosedation; mechanical ventilation; ECMO; ICU; Intensive Care Unit; Critical Care; sedation protocol; analgesia
MeSH Terms: conditions — Respiratory Distress Syndrome; Agnosia; Shock, Cardiogenic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- ECMO patients: Mechanically ventilated adult ICU patients who received ECMO organ support
  Interventions: Other: Not an intervention study
- Healthcare professionals: Doctors, nurses and pharmacists who look after ECMO patients
  Interventions: Other: Not an intervention study
- Non-ECMO: Mechanically ventilated adult ICU patients who did not receive ECMO organ support
  Interventions: Other: Not an intervention study
- ECMO survivors and family: ECMO survivors who have recovered and discharged from hospital. Family of ECMO survivors.
  Interventions: Other: Not an intervention study

INTERVENTIONS:
Other: Not an intervention study — This is not an intervention study

SUMMARY:
Sedation (painkillers and sedative drugs) treats pain, reduces suffering, and helps patients in the intensive care unit (ICU) receiving extracorporeal membrane oxygenation (ECMO) remain comfortable. ECMO is a life support machine that provides oxygen and removes waste gases (carbon dioxide) in very sick patients with severe heart or lung failure. About 300-400 patients per year receive ECMO in the UK. These patients are younger and generally more healthy compared to other critically ill patients. However patients that survive ECMO have long-term health problems. These include anxiety, memory problems, withdrawal from medicines, and mobility issues. These problems issues could all be related to the type and amount of sedation given.

A sedation protocol is a way of guiding healthcare professionals how much sedation is given to patients in ICU. Too much sedation can cause confusion, hallucinations, excessive sleepiness, and longer time in hospital. Too little sedation can cause pain, distress, and also a longer time in hospital. Using a sedation protocol in non-ECMO patients has been shown to reduce these complications.

However, there are no protocols for giving sedation to ECMO patients in research papers. The investigators know healthcare staff find it difficult to manage sedation, and higher amounts of sedation is given to ECMO patients.

Aims:

* To describe current sedation use in ECMO patients in the UK and compare to non-ECMO critically ill patients.
* To develop a sedation protocol for ECMO patients with input from patients, their family, and staff.

Design/methods:

Study 1:

The investigators will study how sedation is used in adult ECMO patients and compare with non-ECMO but critically ill patients in the UK. The investigators will collect information on drug doses and pain and sedation scores. The investigators will also ask ECMO centres if they use a sedation protocol to adjust sedation doses. This information will be helpful for the design of the protocol in study 2.

Study 2:

The investigators will design a sedation protocol with input from patients, family, and staff. The investigators will organise meetings to share experiences and agree on what to include in the protocol that is considered acceptable and safe. The investigators will then assess if the protocol is safe and acceptable with staff outside the co-design group.

Patient and public involvement/engagement:

The investigators received feedback from patients and family members which helped to design this proposal, the lay summary and what to measure in a trial. Patients and family members will continue to help with development of the sedation and trial protocol. They will advise how the investigators should review study findings, and support sharing of results to the public.

Impact/dissemination:

The investigators will share findings through social media, patient charities, research papers and conferences.

DETAILED DESCRIPTION:
Overall Aim and purpose:

• The overall aim is to develop a co-designed analgosedation protocol for adult extracorporeal membrane oxygenation (ECMO) patients and test its acceptability with staff and patients.

Objectives:

Stage 1

* To describe and explore current practices of analgosedation (in terms of opioid and sedative choice, dose and assessment) and use of analgosedation protocols, and sedation holds in ECMO and non-ECMO ICU adult patients.
* To describe patient outcomes (including those recommended by my PPIE advisory group): ICU mortality, ICU length of stay, and delirium incidence.
* To determine clinical equipoise with the direct clinical care team on using a co-designed analgosedation protocol in a feasibility cluster randomised control trial.

Stage 2

• To determine anticipatory acceptability of the co-designed analgosedation protocol.

Study design:

Stage 1: multi-centre observational cohort study reviewing analgosedation practices in UK ECMO centres comparing ECMO to non-ECMO patients The investigators will conduct a prospective multi-centre observational cohort study enrolling UK adult ECMO centres. The investigators aim to recruit all ECMO centres to participate. The investigators are recruiting sites via a well-established national pharmacist and physician ECMO groups. Analgosedation data will be collected for all ECMO patients and a representative sample of non-ECMO ICU patients either in the same unit or another representative ICU in ECMO centres with multiple ICUs. The investigators will collect outcome data to patient discharge from ICU. The investigators will organise meetings with consultant doctors at St Thomas' and Royal Brompton Hospitals to determine clinical equipoise of using a co-designed analgosedation protocol in a feasibility cluster randomised controlled trial versus no protocol.

Data collection:

Data to be collected

Patients:

Sites will record data using a printed case report form. The direct care team will de-identify identifiable patient data before uploading it on to the electronic case report form (e-CRF). The investigators will develop a e-CRF (in collaboration with with King's College London) to collect de-identified patient demographic characteristics, analgosedation management and patient outcomes. Sites will then transfer de-identified data on to the electronic data capture system (REDCap) and lock when completed to ensure patient confidentiality. The investigators will train the direct clinical care team, clinical pharmacists and research nurses at participating sites on data collection. Data collected will include baseline characteristics (age, gender, weight, height, APACHE II score and past medical history), continuous analgosedative (opioid and/or sedative) IV infusion hourly doses (excluding bolus doses), and enteral opioid and sedatives doses during a 5-day observation period documented in the patient medical record. The investigators will also document type and numerical values of pain score, sedation scores (Richmond, Agitation and Sedation Score (RASS)), delirium presence (assessed by Confusion Assessment Method for the Intensive Care Unit, CAM-ICU) and duration during the 5-day collection period Outcome data including ICU length of stay, ECMO duration and ICU mortality will be collected.

Consultant doctors:

The investigators will collect information on the number of consultant doctors who attend the meeting to review clinical equipoise, the total number of consultant doctors employed within each service, and the number of consultant doctors who confirm clinical equipoise.

Data analysis:

Quantitative analysis:

The investigators will calculate the median (interquartile range) of daily (24 hour period) dose of each analgosedation drug. The investigators will convert all opioids (enteral and intravenous) to morphine dose equivalents; benzodiazepines (enteral and intravenous) into midazolam dose equivalents using opioid and benzodiazepine conversion tables. The investigators will calculate median daily dose by dividing the sum of all analgosedation doses received during the data collection period by the number of days of collected data. To compare analgosedation doses and patient outcomes of ECMO versus non-ECMO ICU patients, the investigators will test data for normality and use summary measures for central tendency (mean, median) and variability (standard deviation, interquartile range, minimum, maximum). The investigators will present categorical data as counts (%). Comparisons will be made using parametric t-test or non-parametric Wilcoxon rank sum test depending on data distribution. The investigators will use univariable and multivariable linear regression with a priori selected co-variates to examine the association between patient factors and analgosedation dosing including use of ECMO. Data will be analysed using R Studio.

Stage 2

Study design

The investigators will conduct a mixed methods study to determine anticipatory acceptability of a co-designed protocol using the Theoretical Framework of Acceptability questionnaire informed by the Theoretical Framework of Acceptability (TFA).

Data to be collected

The investigators will develop an interview guide addressing the seven domains (affective attitude, burden, ethnicality, perceived effectiveness, intervention coherence, self-efficacy and opportunity costs) of the TFA to qualitatively assess acceptability of the co-designed protocol. The investigators will administer the TFA Questionnaire at the start of the interview to obtain a quantitative score of acceptability. Interviews will be on-line (each lasting 45 minutes long) using Microsoft Teams, digitally recorded and transcribed by a professional transcription company.

Patients and family (NHS and non-NHS participants)

The investigators will collect data including name, age, contact details, gender, ethnicity, and job status for patients, family taking part.

Healthcare staff (NHS participants)

The investigators will collect data including name, age, contact details, gender, ethnicity, professional role, location of job, length of time in current position, and duration of intensive care career to date for healthcare staff taking part.

Data analysis

Qualitative analysis:

The investigators will use The Framework Method using the TFA concepts as the backbone of the framework. The investigators will dual-code transcripts coding data within the domains of the TFA. The investigators will group and mark codes from the transcripts with one or more short descriptors to organise the raw data. The codes will then be grouped, summarised and categorised according to their meaning, similarities and differences. The investigators will use the data management tool NVivo to support the coding and the analysis of the qualitative data. The investigators will use the consolidated criteria for reporting qualitative studies (COREQ) validated checklist to ensure transparent reporting, rigor and credibility.

Quantitative analysis The investigators will analyse the scores from the TFA questionnaire computing the total mean score of the 7 domains as a single acceptability score.

Following analysis of both qualitative and quantitative datasets, the investigators will integrate both using established methodological triangulation to provide a mixed methods interpretation. This involves comparing both qualitative and quantitative datasets to confirm areas of convergence and divergence in the two datasets. Triangulation will help to increase validity of the research findings and explain research biases. The investigators will integrate findings using a convergence-coding matrix.

ELIGIBILITY:
Stage 1 (multi-centre observational study):

Inclusion Criteria:

1. Aged 18 years and older.
2. Receiving continuous IV infusions of analgosedation (opioids, benzodiazepines, and/or propofol).
3. Receiving ECMO for moderate to severe respiratory failure (PaO2/FiO2 (P/F) ratio <20 kilopascals (kPa)) for ≤ 7 days during the week of recruitment.
4. Non-ECMO ICU patients (control group): must satisfy inclusion criteria 1 and 2, and have received mechanical ventilation for moderate to severe respiratory failure (P/F ratio < 20kPa) for at least 48 hours OR mechanical ventilation for cardiovascular disorder (out of hospital cardiac arrest, following cardiothoracic or transplant surgery or percutaneous coronary intervention or acute heart failure).

Exclusion Criteria:

1. Anticipated length of ICU stay in recruiting centre for less than 24 hours.
2. Withdrawal of life-sustaining treatment in the next 24 hours.

Stage 2 (mixed methods study):

Inclusion Criteria:

1. Healthcare professionals working at one of two ECMO centres (St Thomas' Hospital and Royal Brompton Hospital (part of Guy's and St Thomas' NHS Foundation Trust).
2. ECMO survivors (patients admitted to ICU and survived ECMO organ support) who have returned home, and recovered.
3. Family members of ECMO survivors, whose relative is no longer hospitalised.

Exclusion Criteria:

1. ECMO survivors currently receiving treatment in hospital.
2. ECMO survivors with severe cognitive issues (issues with short-term memory and thinking).
3. ECMO survivors who cannot communicate in English.
4. Non-ECMO survivors and family members.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — All
Study Population: Stage 1: mechanically ventilated adult ICU patients Stage 2: Healthcare professionals (doctors, nurses and pharmacists) with experience caring for ECMO patients. ECMO survivors who have recovered and discharged from hospital, and their family.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
ICU mortality | Through study completion, an average of 1 year
  Death whilst in ICU

OTHER OUTCOMES:
ICU length of stay | Through study completion, an average of 1 year
  Length of stay in tertiary ICU
Delirium | Through study completion, an average of 1 year
  Occurrence of delirium during study period

CONTACTS AND LOCATIONS:
Overall Officials: Louise Rose, PhD, Study Chair — King's College London
Locations (1):
- Guy's and St Thomas' NHS Foundation Trust, London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The King's Open Research Data System (KORDS) at King's College London will be used as a data repository, which will provide long-term storage and access for anonymised data and study protocol at project-end and to support publications. KORDS uses the Figshare data repository platform, providing a simple, self-deposit way for researchers to upload and share their data, and a publicly accessible showcase of datasets from King's research. It supports Open Research, enabling researchers to make datasets discoverable, accessible and citeable. All datasets have a DOI and a structured metadata record so that they can be shared and cited when re-used. Depositing meets the policy requirements of funders for data retention and sharing, and the requirements of many publishers for access to datasets supporting publications.
Supporting Information: Study Protocol
Time Frame: The data will be made available following publication of research findings in peer-reviewed manuscripts and presentation at international conferences.
Access Criteria: Institution access will be needed to access any data. This includes permission to access the specific university and hospital servers. Potential users will require tools including Microsoft Excel and Microsoft Word to access and use the data, which are widely adopted in many institutions and sustainable. The data will be shared via the University repository KORDS but it will not be openly accessible. Requests for access to the data will be handled directly by the research team in line with local policies.
URL: https://www.kcl.ac.uk/researchsupport/managing/preserve

REFERENCES:
- [Background] Rose L, Fitzgerald E, Cook D, Kim S, Steinberg M, Devlin JW, Ashley BJ, Dodek P, Smith O, Poretta K, Lee Y, Burns K, Harvey J, Skrobik Y, Fergusson D, Meade M, Kraguljac A, Burry L, Mehta S; SLEAP Investigators; Canadian Critical Care Trials Group. Clinician perspectives on protocols designed to minimize sedation. J Crit Care. 2015 Apr;30(2):348-52. doi: 10.1016/j.jcrc.2014.10.021. Epub 2014 Oct 30. PMID 25466317
- [Background] Rose RL, Bucknall T. Staff perceptions on the use of a sedation protocol in the intensive care setting. Aust Crit Care. 2004 Nov;17(4):151-9. doi: 10.1016/s1036-7314(04)80020-1. PMID 18038524
- [Background] Shehabi Y, Bellomo R, Kadiman S, Ti LK, Howe B, Reade MC, Khoo TM, Alias A, Wong YL, Mukhopadhyay A, McArthur C, Seppelt I, Webb SA, Green M, Bailey MJ; Sedation Practice in Intensive Care Evaluation (SPICE) Study Investigators and the Australian and New Zealand Intensive Care Society Clinical Trials Group. Sedation Intensity in the First 48 Hours of Mechanical Ventilation and 180-Day Mortality: A Multinational Prospective Longitudinal Cohort Study. Crit Care Med. 2018 Jun;46(6):850-859. doi: 10.1097/CCM.0000000000003071. PMID 29498938
- [Background] Kress JP, Pohlman AS, O'Connor MF, Hall JB. Daily interruption of sedative infusions in critically ill patients undergoing mechanical ventilation. N Engl J Med. 2000 May 18;342(20):1471-7. doi: 10.1056/NEJM200005183422002. PMID 10816184
- [Background] Devlin JW, Skrobik Y, Gelinas C, Needham DM, Slooter AJC, Pandharipande PP, Watson PL, Weinhouse GL, Nunnally ME, Rochwerg B, Balas MC, van den Boogaard M, Bosma KJ, Brummel NE, Chanques G, Denehy L, Drouot X, Fraser GL, Harris JE, Joffe AM, Kho ME, Kress JP, Lanphere JA, McKinley S, Neufeld KJ, Pisani MA, Payen JF, Pun BT, Puntillo KA, Riker RR, Robinson BRH, Shehabi Y, Szumita PM, Winkelman C, Centofanti JE, Price C, Nikayin S, Misak CJ, Flood PD, Kiedrowski K, Alhazzani W. Clinical Practice Guidelines for the Prevention and Management of Pain, Agitation/Sedation, Delirium, Immobility, and Sleep Disruption in Adult Patients in the ICU. Crit Care Med. 2018 Sep;46(9):e825-e873. doi: 10.1097/CCM.0000000000003299. PMID 30113379
- [Background] Ely EW, Shintani A, Truman B, Speroff T, Gordon SM, Harrell FE Jr, Inouye SK, Bernard GR, Dittus RS. Delirium as a predictor of mortality in mechanically ventilated patients in the intensive care unit. JAMA. 2004 Apr 14;291(14):1753-62. doi: 10.1001/jama.291.14.1753. PMID 15082703
- [Background] Remmington C, McKenzie C, Camporota L, Hanks F, Barker M, Sanderson B, Rose L. Analgosedation in extracorporeal membrane oxygenation: a retrospective UK cohort study. Br J Anaesth. 2023 Aug;131(2):e50-e52. doi: 10.1016/j.bja.2023.05.011. Epub 2023 Jun 19. No abstract available. PMID 37344336
- [Background] Grap MJ, Munro CL, Wetzel PA, Best AM, Ketchum JM, Hamilton VA, Arief NY, Pickler R, Sessler CN. Sedation in adults receiving mechanical ventilation: physiological and comfort outcomes. Am J Crit Care. 2012 May;21(3):e53-63; quiz e64. doi: 10.4037/ajcc2012301. PMID 22549581
- [Background] Balzer F, Weiss B, Kumpf O, Treskatsch S, Spies C, Wernecke KD, Krannich A, Kastrup M. Early deep sedation is associated with decreased in-hospital and two-year follow-up survival. Crit Care. 2015 Apr 28;19(1):197. doi: 10.1186/s13054-015-0929-2. PMID 25928417
- [Background] Kamdar BB, Combs MP, Colantuoni E, King LM, Niessen T, Neufeld KJ, Collop NA, Needham DM. The association of sleep quality, delirium, and sedation status with daily participation in physical therapy in the ICU. Crit Care. 2016 Aug 18;19:261. doi: 10.1186/s13054-016-1433-z. PMID 27538536
- [Background] Dzierba AL, Abrams D, Brodie D. Medicating patients during extracorporeal membrane oxygenation: the evidence is building. Crit Care. 2017 Mar 21;21(1):66. doi: 10.1186/s13054-017-1644-y. PMID 28320466
- [Background] Shekar K, Abdul-Aziz MH, Cheng V, Burrows F, Buscher H, Cho YJ, Corley A, Diehl A, Gilder E, Jakob SM, Kim HS, Levkovich BJ, Lim SY, McGuinness S, Parke R, Pellegrino V, Que YA, Reynolds C, Rudham S, Wallis SC, Welch SA, Zacharias D, Fraser JF, Roberts JA. Antimicrobial Exposures in Critically Ill Patients Receiving Extracorporeal Membrane Oxygenation. Am J Respir Crit Care Med. 2023 Mar 15;207(6):704-720. doi: 10.1164/rccm.202207-1393OC. PMID 36215036
- [Background] Shekar K, Fraser JF, Smith MT, Roberts JA. Pharmacokinetic changes in patients receiving extracorporeal membrane oxygenation. J Crit Care. 2012 Dec;27(6):741.e9-18. doi: 10.1016/j.jcrc.2012.02.013. Epub 2012 Apr 18. PMID 22520488
- [Background] Kim M, Mahmood M, Estes LL, Wilson JW, Martin NJ, Marcus JE, Mittal A, O'Connell CR, Shah A. A narrative review on antimicrobial dosing in adult critically ill patients on extracorporeal membrane oxygenation. Crit Care. 2024 Oct 4;28(1):326. doi: 10.1186/s13054-024-05101-z. PMID 39367501
- [Background] Marhong JD, DeBacker J, Viau-Lapointe J, Munshi L, Del Sorbo L, Burry L, Fan E, Mehta S. Sedation and Mobilization During Venovenous Extracorporeal Membrane Oxygenation for Acute Respiratory Failure: An International Survey. Crit Care Med. 2017 Nov;45(11):1893-1899. doi: 10.1097/CCM.0000000000002702. PMID 28863011
- [Background] Dzierba AL, Abrams D, Madahar P, Muir J, Agerstrand C, Brodie D. Current practice and perceptions regarding pain, agitation and delirium management in patients receiving venovenous extracorporeal membrane oxygenation. J Crit Care. 2019 Oct;53:98-106. doi: 10.1016/j.jcrc.2019.05.014. Epub 2019 May 29. PMID 31202165
- [Background] deBacker J, Tamberg E, Munshi L, Burry L, Fan E, Mehta S. Sedation Practice in Extracorporeal Membrane Oxygenation-Treated Patients with Acute Respiratory Distress Syndrome: A Retrospective Study. ASAIO J. 2018 Jul/Aug;64(4):544-551. doi: 10.1097/MAT.0000000000000658. PMID 29045280
- [Background] Brodie D, Bacchetta M. Extracorporeal membrane oxygenation for ARDS in adults. N Engl J Med. 2011 Nov 17;365(20):1905-14. doi: 10.1056/NEJMct1103720. PMID 22087681